CLINICAL TRIAL: NCT06564103
Title: Stratification for Efficacy of Adjuvant FOLFOX Plus Lenvatinib After Liver Transplantation for Hepatocellular Carcinoma in Recurrence Prevention
Brief Title: Stratification for F-L Therapy After LT
Status: Completed | Type: Observational
Sponsor: Xiao Xu (Other)
Responsible Party: Sponsor-Investigator, Xiao Xu, Principal Investigator, Clinical Professor,PHD,MD, Zhejiang University
Organization: Zhejiang University (Other)
Other Study IDs: CT2024-ZJU-OBS10
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Liver Transplantation; Adjuvant FOLFOX Plus Lenvatinib; Machine Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adjuvant FOLFOX plus lenvatinib therapy group
- non-adjuvant therapy group

INTERVENTIONS:
Combination Product:
  Groups: non-adjuvant therapy group

SUMMARY:
Objective: To stratify recipients who underwent adjuvant FOLFOX plus lenvatinib (F-L) therapy following liver transplantation (LT) for hepatocellular carcinoma and provide guidance for clinical adjuvant therapy.

Methods: Liver recipients in the Shulan (Hangzhou) Hospital from January, 2017 to December, 2021, including 106 in the F-L therapy group and 229 in the non-adjuvant (N-A) therapy group were included in the analysis. A 1:1 propensity score matching (PSM) analysis was performed to minimize group imbalances. Disease-free survival (DFS) and overall survival (OS) were compared among recipients. Radiomics features that demonstrated predictive value for recurrence were employed, either independently or in conjunction with prognostic clinical features, to formulate predictive models. The combined model was used to perform further subgroup analysis for recipients in the F-L therapy group.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilling the Hangzhou criteria or exceeding the Hangzhou criteria with type 1 or 2 portal vein tumor thrombus (PVTT) before LT

Exclusion Criteria:

* 1) individuals less than 18 years old; 2) individuals with malignancies other than HCC; 3) individuals who survived less than 30 days after LT; and 4) individuals who lacked important prognostic variables, such as contrast-enhanced CT imaging information one month before transplantation, preoperative alpha-fetoprotein (AFP) levels, and tumor differentiation data

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recipients at Shulan (Hangzhou) Hospital from January 2017 to December 2021 were included in the analysis, which comprised 106 recipients in the F-L therapy group and 229 non-adjuvant (N-A) therapy group recipients.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
The disease-free survival rate was evaluated by follow-up investigation and outpatient review | 1-5 years

SECONDARY OUTCOMES:
The overall survival rate was evaluated by follow-up investigation and outpatient review | 1-5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University school of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided